CLINICAL TRIAL: NCT04383574
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial, to Evaluate Safety and Immunogenicity of Inactivated SARS-CoV-2 Vaccine (Vero Cell), in Healthy Elderly Aged 60 Years and Above
Brief Title: Safety and Immunogenicity Study of Inactivated Vaccine for Prevention of SARS-CoV-2 Infection(COVID-19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-nCOV-1002
Record Dates: First submitted 2020-05-09; First posted 2020-05-12 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Vaccine-medium dosage (Experimental): 24 participants in medium-dosage group in phase Ⅰ will receive two doses of primary immunization according to the immunization schedule of day 0, 28 and will receive 1 dose of booster immunization 1 year after primary immunization; 100 participants in medium-dosage group in phase Ⅱ will receive two doses of primary immunization according to the immunization schedule of day 0,28 ,1 dose of booster immunization 6 months after primary immunization(the third dose ) and the second booster dose (the fourth dose) 1 year after the second dose.
  Interventions: Biological: Two doses of medium dosage inactivated SARS-CoV-2 vaccine at the schedule of day 0,28
- Experimental Vaccine-high dosage (Experimental): 24 participants in high-dosage group in phase Ⅰ will receive two doses of primary immunization according to the immunization schedule of day 0, 28 and will receive 1 dose of booster immunization 1 year after primary immunization; 100 participants in high-dosage group in phase Ⅱ will receive two doses of primary immunization according to the immunization schedule of day 0,28 ,1 dose of booster immunization 6 months after primary immunization(the third dose) and the second booster dose (fourth dose) 1 year after the second dose .
  Interventions: Biological: Two doses of high dosage inactivated SARS-CoV-2 vaccine at the schedule of day 0,28
- Placebo (Placebo Comparator): 24 participants including 12 at medium dosage stage and 12 at high dosage in phase Ⅰ will receive two doses of placebo according to the immunization schedule of day 0, 28 and will receive 1 dose of booster immunization 1 year after primary immunization; 50 participants in phase Ⅱ will receive two doses of primary immunization according to the immunization schedule of day 0,28 and will receive 1 dose of booster immunization 6 months after primary immunization.
  Interventions: Biological: Two doses of placebo at the schedule of day 0,28
- Experimental Vaccine-low dosage (Experimental): 100 participants at low dosage stage in phase Ⅱ will receive two doses of primary immunization according to the immunization schedule of day 0,28 and will receive 1 dose of booster immunization 6 months after primary immunization.
  Interventions: Biological: Two doses of low dosage inactivated SARS-CoV-2 vaccine at the schedule of day 0,28

INTERVENTIONS:
Biological: Two doses of medium dosage inactivated SARS-CoV-2 vaccine at the schedule of day 0,28 — The inactivated SARS-CoV-2 vaccine was manufactured by Sinovac Research & Development Co., Ltd..Two doses of medium dosage (600SU/0.5ml) experimental vaccine at the schedule of day 0,28,and one dose of booster immunization(the third dose) with medium dosage (600SU/0.5ml) experimental vaccine 1 year after primary immunization at the schedule of day 0,28 in phaseⅠand 6 months after primary immunization at the schedule of day 0,28 in phase Ⅱ.And the second booster dose (the fourth dose) 1 year after the second dose.
  Arms: Experimental Vaccine-medium dosage
Biological: Two doses of high dosage inactivated SARS-CoV-2 vaccine at the schedule of day 0,28 — The inactivated SARS-CoV-2 vaccine was manufactured by Sinovac Research & Development Co., Ltd..Two doses of high dosage (1200SU/0.5ml) experimental vaccine at the schedule of day 0,28,and one dose of booster immunization(the third dose) with medium dosage (1200SU/0.5ml) experimental vaccine 1 year after primary immunization at the schedule of day 0,28 in phaseⅠand 6 months after primary immunization at the schedule of day 0,28 in phase Ⅱ.And the second booster dose (the fourth dose) 1 year after the second dose.
  Arms: Experimental Vaccine-high dosage
Biological: Two doses of placebo at the schedule of day 0,28 — The placebo was manufactured by Sinovac Research & Development Co., Ltd., Two doses of placebo at the schedule of day 0,28,and one dose of booster immunization with placebo 1 year after primary immunization at the schedule of day 0,28 in phaseⅠand 6 months after primary immunization at the schedule of day 0,28 in phase Ⅱ.
  Arms: Placebo
Biological: Two doses of low dosage inactivated SARS-CoV-2 vaccine at the schedule of day 0,28 — The inactivated SARS-CoV-2 vaccine was manufactured by Sinovac Research & Development Co., Ltd..Two doses of low dosage (300SU/0.5ml)experimental vaccine at the schedule of day 0,28,and one dose of booster immunization with low dosage (300SU/0.5ml) experimental vaccine 6 months after primary immunization at the schedule of day 0,28 in phase Ⅱ.
  Arms: Experimental Vaccine-low dosage

SUMMARY:
This study is a randomized, double-blinded, and placebo controlled phase 1&2 clinical trial of the SARS-CoV-2 inactivated vaccine manufactured by Sinovac Life Sciences Co. , Ltd. The purpose of this study is to evaluate the safety and immunogenicity of the experimental vaccine in healthy elderly aged 60 years and above.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, single-center, placebo-controlled phase 1&2 clinical trial in healthy elderly aged 60 years and above. The experimental vaccine and placebo were both manufactured by Sinovac Life Sciences Co. , Ltd. A total of 422 subjects will be enrolled, with 72 in phase 1 and 350 in phase 2. 72 Subjects with 36 in medium-dosage group and 36 in high-dosage group in phase 1 will receive two doses of primary immunization according to the immunization schedule of day 0, 28 and the subjects at each dosage group will be assigned in a 2:1 ratio to receive investigational vaccine or placebo respectively.All enrolled subjects will receive 1 dose of booster immunization 1 year after primary immunization.350 Subjects in phase 2 will receive two doses of primary immunization according to the immunization schedule of day 0,28,the subjects will be assigned in a ratio of 2:2:2:1 to receive the low dosage, medium dosage, high dosage vaccine, or placebo. All enrolled subjects will received 1 dose of booster immunization(the third dose ) 6 months after primary immunization.And subjects in medium-dosage group and high -dosage group will receive the second booster dose (the fourth dose) 1 year after the second dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥60 years;
* Be able to understand and sign the informed consent voluntarily;
* Provide legal identification;

Exclusion Criteria:

* Travel / residence history of Wuhan city and surrounding areas or other communities with case reports within 14 days prior to the enrolment;
* Contact with SARS-CoV-2 infected persons (positive for nucleic acid detection) within 14 days prior to the enrolment;
* Contact patients with fever or respiratory symptoms from Wuhan city and surrounding areas, or from communities with case reports within 14 days prior to the enrolment;
* Two or more cases of fever and / or respiratory symptoms in a small contact area of subjects, such as family, office, school class or other places within 14 days prior to the enrolment;
* History of SARS;
* History of SARS-CoV-2 infection;
* History of asthma, allergy to vaccines or vaccine ingredients, and serious adverse reactions to vaccines, such as urticaria, dyspnea, angioneuroedema;
* Congenital malformation or developmental disorder, genetic defect, severe malnutrition, etc;
* Autoimmune disease or immunodeficiency / immunosuppression;
* Serious chronic disease, serious cardiovascular disease, hypertension and diabetes that cannot be controlled by drugs, hepatorenal disease, malignant tumor, etc;
* Serious nervous system disease (epilepsy, convulsion or convulsion) or psychosis;
* Thyroid disease or history of thyroidectomy, asplenia, functional asplenia, asplenia or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute non-complicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* Long history of alcohol or drug abuse;
* Receipt of blood products in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Acute diseases or acute exacerbation of chronic diseases in the past 7 days;
* Axillary temperature >37.0°C;
* According to the investigator's judgment, the subject has any other factors that are not suitable for the clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Safety index-incidence of adverse reactions | Day 0-28 after each dose vaccination
  Incidence of adverse reactions after each dose vaccination
Immunogenicity index-seroconversion rates of neutralizing antibody | 28 days after the second dose vaccination
  The seroconversion rate of neutralizing antibody 28 days after the second dose vaccination.

SECONDARY OUTCOMES:
Safety index-incidence rate of adverse reactions | within 7 days after each dose vaccination
  Incidence rate of adverse reactions within 7 days after each dose vaccination
Safety index-incidence rate of serious adverse events in phase Ⅰ | From the beginning of the vaccination to 6 months after the booster immunization
  Incidence rate of SAEs from the beginning of the vaccination to 6 months after the booster immunization in phase Ⅰ
Safety index-incidence rate of serious adverse events in phase Ⅱ | From the beginning of the vaccination to 12 months after the booster immunization vaccination
  Incidence rate of SAEs from the beginning of the vaccination to 12 months after the booster immunization vaccination in phase Ⅱ
Immunogenicity index-seropositive rate, GMT, and GMI of neutralizing antibodies | 28 days after the second dose vaccination
  The seropositive rate, GMT, and GMI of neutralizing antibodies 28 days after the second dose vaccination;
Immunogenicity index-seroconversion rate, seropositive rate, GMT, and GMI in phase Ⅰ | 28 days after the first dose vaccination in phase Ⅰ
  The seroconversion rate, seropositive rate, GMT, and GMI 28 days after the first dose vaccination in phase Ⅰ

OTHER OUTCOMES:
Immunogenicity index -seropositive rate and GMT of neutralizing antibodies | 6 months after the second dose vaccination
  The seropositive rate and GMT 6 months after the second dose vaccination
Immunogenicity index -seropositive rate and GMT of neutralizing antibodies in phase Ⅰ | 12 months after the second dose vaccination
  The seropositive rate and GMT 12 months after the second dose vaccination in phase Ⅰ
Immunogenicity index -seropositive rate, GMT, and GMI of neutralizing antibodies | 28 days after the booster vaccination
  The seropositive rate, GMT, and GMI 28 days after the booster vaccination in phase Ⅰ
Immunogenicity index -seropositive rate, GMT of neutralizing antibodies in phase Ⅱ | 7 days (or 14 days) and 28 days after the booster vaccination
  The seropositive rate, GMT, and GMI 7 days (or 14 days) and 28 days after the booster vaccination in phase Ⅱ
Immunogenicity index -seropositive rate and GMT of neutralizing antibodies | 6 months after the booster vaccination
  The seropositive rate and GMT 6 months after the booster vaccination
Immunogenicity index -seropositive rate and GMT of neutralizing antibodies in phase Ⅱ | 12 months after the booster vaccination
  The seropositive rate and GMT 12 months after the booster vaccination in phase Ⅱ
Immunogenicity index-seropositive rate,GMT and GMI of neutralizing antibodies | 14 days after the fourth dose
  The seropositive rate, GMT and GMI of neutralizing antibody against CZ, Delta and Omicron antigens 14 days after the fourth dose.
Immunogenicity index-Seropositive rate and GMTof neutralizing antibodies | 6 months after the fourth dose
  The seropositive rate and GMT of neutralizing antibody against Delta and Omicron antigens 6 months after the fourth dose.

CONTACTS AND LOCATIONS:
Overall Officials: Yuliang Zhao, Master, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Renqiu City Center for Disease Control and Prevention, Renqiu, Hebei, China

REFERENCES:
- [Derived] Xin Q, Wu Q, Chen X, Han B, Chu K, Song Y, Jin H, Chen P, Lu W, Yang T, Li M, Zhao Y, Pan H, Yu H, Wang L. Six-month follow-up of a booster dose of CoronaVac in two single-centre phase 2 clinical trials. Nat Commun. 2022 Jun 3;13(1):3100. doi: 10.1038/s41467-022-30864-w. PMID 35660738
- [Derived] Zeng G, Wu Q, Pan H, Li M, Yang J, Wang L, Wu Z, Jiang D, Deng X, Chu K, Zheng W, Wang L, Lu W, Han B, Zhao Y, Zhu F, Yu H, Yin W. Immunogenicity and safety of a third dose of CoronaVac, and immune persistence of a two-dose schedule, in healthy adults: interim results from two single-centre, double-blind, randomised, placebo-controlled phase 2 clinical trials. Lancet Infect Dis. 2022 Apr;22(4):483-495. doi: 10.1016/S1473-3099(21)00681-2. Epub 2021 Dec 8. PMID 34890537
- [Derived] Wu Z, Hu Y, Xu M, Chen Z, Yang W, Jiang Z, Li M, Jin H, Cui G, Chen P, Wang L, Zhao G, Ding Y, Zhao Y, Yin W. Safety, tolerability, and immunogenicity of an inactivated SARS-CoV-2 vaccine (CoronaVac) in healthy adults aged 60 years and older: a randomised, double-blind, placebo-controlled, phase 1/2 clinical trial. Lancet Infect Dis. 2021 Jun;21(6):803-812. doi: 10.1016/S1473-3099(20)30987-7. Epub 2021 Feb 3. PMID 33548194